CLINICAL TRIAL: NCT01684007
Title: Clinical Outcomes After Implantation of the AcrySof® IQ ReSTOR® +2.5 D Multifocal Intraocular Lens (MIOL) in the Dominant Eye and Randomization of the AcrySof® IQ ReSTOR® +2.5 D or +3.0 D MIOL in the Fellow Eye
Brief Title: A Clinical Outcome Study of Two Multifocal Intraocular Lenses (IOL) in Cataract Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M-12-007
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-05

CONDITIONS: Cataracts
Keywords: Intraocular lens; Multifocal intraocular lens (MIOL)
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bilateral (Experimental): AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0], bilateral implantation
  Interventions: Device: AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0]
- Contralateral (Active Comparator): AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0] and AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL Model SN6AD1, contralateral implantation
  Interventions: Device: AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0]; Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL Model SN6AD1

INTERVENTIONS:
Device: AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0] — Multifocal IOL with extended secondary focal point implanted for long-term use over the lifetime of the cataract patient
Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL Model SN6AD1 — Multifocal IOL implanted for long-term use over the lifetime of the cataract patient
  Arms: Contralateral

SUMMARY:
The purpose of this study is to compare AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL in both eyes (bilateral implantation) to AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL in the dominant eye with AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL in the fellow eye (contralateral implantation) at Month 3 following the second eye surgery.

DETAILED DESCRIPTION:
Each subject will complete a preoperative examination of both eyes, implantation of IOL at the operative visit for each eye, and up to 4 postoperative visits (each eye examined at Day 1-2, with binocular visits at Day 30 and Day 90 after the second implantation). The second implantation will occur between 1 and 45 days of the first. If the first eye is not implanted during surgery, the second eye is not eligible. lf both eyes are not implanted with the assigned IOL, the subject will be followed for safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand and sign informed consent, and attend postoperative examinations per protocol schedule;
* Requires cataract extraction followed by posterior intraocular lens implantation used as an on-label procedure in both eyes;
* Willing to have second eye surgery within 45 days of first eye surgery;
* Expected postoperative astigmatism < 1.0 D in both eyes, as measured by keratometry;
* Free of severe diseases(s)/condition(s) listed in the Warnings and Precautions section of the package inserts;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Refractive lens exchange (monocular DCVA of worse than 20/20, or ≥ 0.06 logMAR). This exclusion did not apply to binocular (OU) measurement;
* Significant irregular corneal astigmatism as demonstrated by corneal topography;
* Severe degenerative visual disorders;
* Previous corneal surgery;
* Amblyopia;
* Planned multiple procedures, including LRI, LASIK, etc, during surgery or the course of the study;
* History of corneal disease;
* Severe diabetic retinopathy;
* History of retinal detachment;
* Severe conditions or acute or chronic diseases or illnesses that, per investigator's clinical judgment, would increase the operative risk or confound the results of the study;
* Pregnant or planning pregnancy during course of study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magda Michna, PhD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 8 investigative sites located outside the USA, including Argentina (1), Chile (1), Germany (2), Netherlands (2), and Spain (2).
Pre-assignment Details: Of the 112 subjects enrolled, 9 were discontinued prior to randomization as screen failures. This reporting group includes all implanted subjects (103).
Groups:
- Bilateral: AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL, bilateral implantation
- Contralateral: AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL and AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL, contralateral implantation
Period: Overall Study
Arm/Group | Bilateral | Contralateral
Started | 53 | 50
Completed | 53 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all implanted subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bilateral | Contralateral | Total
Number analyzed (Participants) | 53 | 50 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (7.9) | 65.9 (10.1) | 66.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 31 | 66
  Male | 18 | 19 | 37
Region of Enrollment [Number; unit: participants]
  Germany | 13 | 13 | 26
  Netherlands | 12 | 9 | 21
  Spain | 11 | 12 | 23
  Argentina | 7 | 7 | 14
  Chile | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Binocular Distance Corrected Visual Acuity (logMAR) - Intermediate (60 cm)
Description: Visual acuity (VA) was tested binocularly (both eyes together) using the manifest refraction adjusted for optical infinity and the hand-held, 100% contrast, Early Treatment Diabetic Retinopathy Study (ETDRS) chart set at 60 centimeters (cm) on the nearpoint rod. VA was measured in logarithm minimum angle of resolution (logMAR) increments, with 0.1 logMAR corresponding to 5 letters, or 1 line, on the ETDRS chart. A lower logMAR value denotes better visual acuity.
Time Frame: Day 90 from second eye implantation
Population: This analysis population includes all subjects with both eyes implanted.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bilateral | Contralateral
Number analyzed (Participants) | 53 | 50
logMAR | 0.13 (0.148) | 0.09 (0.133)

2. Secondary Outcome: Binocular Distance Corrected Visual Acuity (logMAR) - Near (40 cm)
Description: VA was tested binocularly using the manifest refraction adjusted for optical infinity and the hand-held, 100% contrast, ETDRS chart set at 40 cm on the nearpoint rod. VA was measured in logMAR increments, with 0.1 logMAR corresponding to 5 letters, or 1 line, on the ETDRS chart. A lower logMAR value denotes better visual acuity.
Time Frame: Day 90 from second eye implantation
Population: This analysis population includes all subjects with both eyes implanted.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bilateral | Contralateral
Number analyzed (Participants) | 53 | 50
logMAR | 0.26 (0.158) | 0.10 (0.134)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (Nov2012-Aug2013). This analysis population includes all participants with attempted IOL implantation (successful or aborted after contact with the eye).
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical sign, whether or not related to the medical device. AEs were collected as solicited comments and as observations by the study Investigator as outlined in the protocol.
Arm/Group | Bilateral | Contralateral
Serious Adverse Events (participants affected / at risk) | 0/53 | 2/50
Other Adverse Events (participants affected / at risk) | 3/53 | 3/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bilateral (N=53) | Contralateral (N=50)
Vertigo (Ear and labyrinth disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bilateral (N=53) | Contralateral (N=50)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.